CLINICAL TRIAL: NCT01654328
Title: Oral Versus Intravenous Hydration to Prevent Contrast Induced Nephropathy
Acronym: INOVATIO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow inclusion
Sponsor: Prof. Dr. J. Wetzels (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. J. Wetzels, Clinical Professor, Radboud University Medical Center
Organization: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL nr.: 40730.091.12
Record Dates: First submitted 2012-07-21; First posted 2012-07-31 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Radiographic Contrast Agent Nephropathy
Keywords: contrast media; kidney injury; hydration
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: sodium chloride tablets (Experimental): Arm A: sodium chloride 1g/10kg of body weight /day per os on day -2 and -1 before contrast exposure. With a maximum dose of 10 gram sodium chloride a day.
  Interventions: Drug: Sodium chloride tablets
- B: isotonic saline intravenously (Active Comparator): Sodium chloride solution (isotonic saline (NaCl 0.9%) total 1000ml in 4 hrs or (in case of heart failure or severe renal failure) 12 hrs before and in 4 or in 12 hrs after contrast administration.
  Interventions: Drug: Isotonic saline intravenously

INTERVENTIONS:
Drug: Sodium chloride tablets — sodium chloride 1g/10kg of body weight /day per os on day -2 and -1 before contrast exposure. With a maximum dose of 10 gram sodium chloride a day.
  Arms: Arm A: sodium chloride tablets
Drug: Isotonic saline intravenously — isotonic saline (Nacl 0.9%) total 1000ml in 4 hrs or (in case of heart failure or severe renal failure) 12 hrs before and in 4 or in 12 hrs after contrast administration.
  Arms: B: isotonic saline intravenously

SUMMARY:
The purpose of this study is to investigate if home-hydration is a non inferior alternative for in-hospital hydration in the prevention of Contrast Induced Nephropathy in high risk patients.

DETAILED DESCRIPTION:
Rationale: Iodinated contrast media are regularly used in diagnostic and interventional procedures. The intravascular use of these contrast media can cause acute kidney injury (Contrast Induced Nephropathy). Contrast Induced Nephropathy is associated with increased morbidity and mortality. There are no treatment options, therefore preventive measures should be taken. Volume expansion reduces the risk of Contrast Induced Nephropathy. Current guidelines for the prevention of Contrast-Induced Nephropathy advise that high risk patients be admitted for hydration with intravenous normal saline for a period of 8-24 hours. This proposal evaluates an alternative method of hydration; home hydration with salt tablets.

Objective: To investigate if home-hydration is a non inferior alternative for in-hospital hydration in the prevention of Contrast Induced Nephropathy in high risk patients.

Study design: multi-centre randomized controlled trial.

Study population: Adult patients > 18 years undergoing an elective procedure involving intravascular administration of iodinated contrast media and at high risk for the development of Contrast Induced Nephropathy (as defined by guideline criteria).

Intervention: Arm A: sodium chloride 1g/10kg of body weight/day per os on day -2 and -1 before contrast exposure. With a maximum dose of 10 gram sodium chloride a day.

Arm B: Nacl 0.9% total 1000ml in 4 hrs or (in case of heart failure or severe renal failure) 12 hrs before and in 4 or in 12 hrs after contrast administration.

Main study parameters/endpoints: The incidence of Contrast Induced Nephropathy, effect on the need for hospitalisation, patient satisfaction.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients who are randomized for home hydration will receive salt tablets and start 48 hrs before the procedure. The risk of taking salt tablets is low, there are some reports of nausea. Because the investigators exclude patients who have decompensated heart failure the use of these amounts of salt is considered safe and the investigators do not expect signs of overhydration. The investigators monitor this by a telephone consult, 24 hours after the intake of the first tablets. Body weight and intake of tablets will be monitored. Before contrast administration a blood and urine sample will be taken.

Patients who are randomized for intravenous hydration will be admitted and will receive standard treatment for high risk patients with the addition of one blood and urine sample taken before contrast administration.

In all patients 48-72 hours after contrast administration a blood sample is taken to check for the development of CIN, this is standard treatment according to the guidelines.

The investigators will ask all patients to fill in a questionnaire on patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years undergoing an elective procedure involving intravascular administration of iodinated contrast media
* high risk for the development of Contrast Induced Nephropathy (as defined by guideline criteria

Exclusion Criteria:

* Age < 18.
* Low risk for the development of CIN, therefore no need for hydration
* Emergency contrast procedure.
* Overt signs of overhydration; orthopnea or pulmonal rales at the time of the first consult.

Double or triple diuretic use for pre-existing heart failure. Severe heart failure, in which case salt load is not safe (physician decision) Severe renal failure (CKD stage V eGFR < 15ml/min/1.73m2) Multiple Myeloma. Repeated contrast exposure < 2 weeks Unstable serum creatinine > 25% change < 6 weeks The inability to provide written informed consent. Participation in another intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be change in the creatinine concentration between the 48-72 hours creatinine levels and the baseline levels, expressed as ratio. | 48-72 hours after contrast administration

SECONDARY OUTCOMES:
we will evaluate the incidence of contrast nephropathy in the groups defined as a rise in serum creatinine of ≥25% or ≥44umol/L 48-72 hours after contrast administration | 48-72 hours after contrast administration
patient satisfaction. | up to 1 week after intervention
  patient satisfacation will be evaluated using a questionnaire
the incidence of adverse events | up to 1 week after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jack Wetzels, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands